CLINICAL TRIAL: NCT04021147
Title: Effect of Brain Training Through Visual Mirror Feedback, Action Observation Training and Motor Imagery on Orofacial Sensorimotor Variables in Asymptomatic Subjects: A Single-blind Randomized Controlled Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: uammadrid9
Record Dates: First submitted 2019-07-08; First posted 2019-07-16 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Exercise; Pain
Keywords: Motor Imagery; Action observation; Visual mirror feedback; Pain pressure thresholds
MeSH Terms: conditions — Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Action Observation (Experimental)
  Interventions: Behavioral: Exercise plus action observation
- Motor Imagery (Experimental)
  Interventions: Behavioral: Exercise plus motor imagery
- Visual mirror feedback (Experimental)
  Interventions: Behavioral: Exercise plus visual mirror feedback
- Orofacial exercise (Active Comparator)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise plus action observation — Orofacial exercise plus action observation (video) of the same exercise
  Arms: Action Observation
Behavioral: Exercise plus motor imagery — Orofacial exercise plus motor imagery of the same exercise
  Arms: Motor Imagery
Behavioral: Exercise plus visual mirror feedback — Exercise plus visual mirror feedback
  Arms: Visual mirror feedback
Behavioral: Exercise — Orofacial exercises
  Arms: Orofacial exercise

SUMMARY:
The main objective of the present study was to evaluate the effects of action observation (AO), visual mirror feedback (VMF), motor imagery (MI) combined with an orofacial exercise program in asymptomatic subjects.

ELIGIBILITY:
Inclusion Criteria:

1. healthy individuals with no pain
2. aged between 18 and 65 years
3. subjects with correct masticatory function and labial and lingual mobility

Exclusion Criteria:

1. individuals who presented systemic, cardiorespiratory, central nervous system or rheumatic diseases, or those who presented any musculoskeletal or craniocervical pathology
2. underage individuals
3. individuals with orofacial pain or temporomandibular disorders at the time of the study; (d) subjects' complaint of toothache or tenderness to percussion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2019-08-10 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Pain pressure thresholds (PPTs) | Change from baseline and immediately post-intervention
  PPT is defined as the minimal amount of pressure where a sense of pressure first changes to pain. The mechanical pressure algometer (Force Ten TM FDX Digital Force Gage) used in this study consisted of a round rubber disk (area, 1 cm2) attached to a pressure (force) gauge. The gauge displays values in kilograms but, because the surface of the rubber tip is 1 cm2, the readings are expressed in kg/cm2. The range of values of the pressure algometer is 0 to 10 kg, with 0.1-kg divisions. The pressure was applied at a rate of 0.31 kg/second (Chesterton et al. 2007). Chesterton et al. (2007) have shown that the reliability of pressure algometry is as high as [ICC=0.91 (95% confidence interval, CI 0.82-0.97)].
Lingual muscle endurance | Change from baseline and immediately post-intervention
  Lingual muscle endurance was assessed using the Iowa Oral Performance Instrument (IOPI) (Adams et al. 2015). The measurement of muscular endurance was carried out by placing a plastic bulb with oblong air content on the hard palate, posterior to the central incisor teeth. The participants were asked to elevate the lingual (through anterior and posterior lingual region) to press the instrument with the maximum possible force for 3 seconds, while monitoring the force exerted, quantified in Newtons. Adams et al. (2015) found moderate to strong reliability for anterior (ICC: 0.58-0.77) and posterior (ICC 0.77-0.84) tongue strength.

SECONDARY OUTCOMES:
Maximal mouth opening (MMO) | Change from baseline and immediately post-intervention
  The craniomandibular scale was used to assess the MMO. It was held with the right hand and the left hand was placed on the forehead to maintain the participant's neutral position. The following verbal command was given: "open your mouth as wide as you can without moving your head". The assessor placed the scale on the incisal edge of the maxillary central incisor that was most vertically oriented, measured vertically to the labioincisal edge of the opposing mandibular incisor, and recorded this as the MMO measurement. Beltran-Alacreu et al. (2014) showed that reliability for MMO was good (inter-rater, ICC= 0.95-0.96; intra-rater, ICC= 0.95-0.96). Zawawi et al. (2003) found that the normal range of mouth opening in women is 40-57 mm and 42-68 mm in men
Lingual extensibility | Change from baseline and immediately post-intervention
  This variable consists of measuring the tongue in centimeters, from the chin to the lingual vertex. Through the use of a lingual depressor, located in the midface sagittal axis at the height of the chin, the subject was asked for a maximum lingual protrusion, extending his tongue as far as possible, indicating that route on the lingual depressor and then measuring that distance. The mean obtained from two measurements was recorded.
Ability to generate mental motor images | Change from baseline and immediately post-intervention
  Movement imagery questionnaire-revised (MIQ-R) is an 8-item self-report inventory and was used to assess visual and kinesthetic motor imagery ability. Four different movements are included in MIQ-R and it is comprised of four visual and four kinesthetic items. For each item, participants read a description of the movement. They then physically perform the movement and were instructed to re-assume the starting position after finishing the movement and before performing the mental task, imaging the movement visually or kinesthetically. Then, each participant rated the ease or difficulty of generating that image on a 7-point scale in which 7 indicates "very easy to see/feel" and 1 "very difficult to see/feel. The internal consistencies of the MIQ-R have been consistently adequate with Cronbach's α coefficients ranging above 0.84 for the total scale, 0.80 for de visual subscale and 0.84 for the kinesthetic subscale (Campos and González 2010).

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided